CLINICAL TRIAL: NCT01819155
Title: Assessment of the Immunogenicity and Safety of an MF59™- Adjuvanted Trivalent Influenza Vaccine and a Non-adjuvanted Trivalent Influenza Vaccine Among Children in Senegal
Brief Title: Immunogenicity and Safety Trial of Adjuvanted and Non-adjuvanted Trivalent Influenza Vaccine in Tropical Africa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Institut de Recherche pour le Developpement (Other Government); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MF59-TIV-SEN-01
Record Dates: First submitted 2013-03-22; First posted 2013-03-27 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-06

CONDITIONS: Influenza
Keywords: influenza; influenza vaccine; immunogenicity; Africa; Senegal
MeSH Terms: conditions — Influenza, Human | interventions — fluad vaccine; vaxigrip; Sodium Chloride; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- adjTIV (Experimental): Children randomized to receive adjTIV
  Interventions: Biological: Adjuvanted seasonal trivalent inactivated influenza vaccine
- TIV (Experimental): Children randomized to receive TIV
  Interventions: Biological: Seasonal trivalent inactivated influenza vaccine
- Placebo (Placebo Comparator): Children randomized to receive Placebo
  Interventions: Biological: Saline (bacteriostatic 0.9% sodium chloride for injection)

INTERVENTIONS:
Biological: Adjuvanted seasonal trivalent inactivated influenza vaccine
  Other Names: Fluad
  Arms: adjTIV
Biological: Seasonal trivalent inactivated influenza vaccine
  Other Names: VaxiGrip
  Arms: TIV
Biological: Saline (bacteriostatic 0.9% sodium chloride for injection)
  Arms: Placebo

SUMMARY:
This study will provide the Senegal Ministry of Health with data on the safety and immunogenicity of adjuvanted trivalent inactivated influenza vaccine (adjTIV) and full-dose seasonal non-adjuvanted trivalent inactivated influenza vaccine (TIV) in children. This data will inform future policy considerations for influenza vaccine. The study is not powered to detect significant differences between vaccines or groups, and no hypotheses are to be tested; therefore, immunogenicity and safety objectives are to be analyzed descriptively.

DETAILED DESCRIPTION:
The is a phase 2b, single-center, randomized, observer-blind, parallel group, placebo-controlled trial of the immunogenicity and safety of adjTIV and seasonal TIV among healthy children aged 6 months through 71 months in the town of Niakhar, Senegal. A total of 300 healthy children will be randomized in a 2:2:1 ratio of adjTIV to TIV to placebo. Each child will receive two doses of one of the three study vaccines, with each dose given 28 days apart. Each child will be followed closely for safety after each dose for the period from one month post-dose two to 3 months post-dose two. For determination of immune response to vaccination or background influenza infection, 3 mL of blood will be obtained at three time points: pre-vaccination, 28 days post-dose one (prior to receipt of dose two), and at 28 days post-dose two. Serum anti-influenza antibodies produced against virus strains contained in the vaccine will be detected using hemagglutination inhibition assay.

ELIGIBILITY:
Inclusion Criteria:

* A male or female child at least 6 months of age and under 6 years of age (has not yet reached 72 months of age) at the enrollment visit.
* Free of obvious health problems, as established by the medical history and screening evaluations, including physical examination.
* Subject's parent or legal guardian is willing to provide written informed consent prior to the subject's first study vaccination.

Exclusion Criteria:

* Known hypersensitivity to any component in adjTIV or TIV (which include egg protein) or placebo.
* Receipt of any non-study vaccine within two weeks prior to enrollment or refusal to postpone receipt of such vaccines until after the Day 56 visit.
* Previous receipt of any influenza vaccine.
* Hypersensitivity after previous administration of any vaccine.
* Acute illness accompanied by a body temperature of 37.5°C or greater (axillary measurement) within 14 days of enrollment visit. (Enrollment and administration of adjTIV, TIV, or placebo should be postponed until at least 14 days after recovery. Minor illnesses, such as mild upper respiratory infection, with an axillary temperature of <37.5°C, are not reason for exclusion or postponing study vaccination.)
* Any condition that, in the opinion of the investigator, would pose a health risk to the participant if he/she participates in the study or would interfere with the evaluation of the study objectives.

Ages: 6 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 296 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Immunogenicity of adjTIV | 28 days post-dose 2
  serum hemagglutination-inhibition antibodies
Immunogenicity of TIV | 28 days post-dose 2
  serum hemagglutination-inhibition antibodies

SECONDARY OUTCOMES:
Adverse events | through three months post-dose 2

CONTACTS AND LOCATIONS:
Overall Officials: Aldiouma Diallo, MD, Principal Investigator — Institut de Recherche pour le Developpement; John C Victor, PhD, MPH, Study Director — PATH
Locations (1):
- Institut de Recherche pour le Développement, Niakhar, Senegal

REFERENCES:
- [Derived] Diallo A, Victor JC, Feser J, Ortiz JR, Kanesa-Thasan N, Ndiaye M, Diarra B, Cheikh S, Diene D, Ndiaye T, Ndiaye A, Lafond KE, Widdowson MA, Neuzil KM. Immunogenicity and safety of MF59-adjuvanted and full-dose unadjuvanted trivalent inactivated influenza vaccines among vaccine-naive children in a randomized clinical trial in rural Senegal. Vaccine. 2018 Oct 15;36(43):6424-6432. doi: 10.1016/j.vaccine.2018.08.032. Epub 2018 Sep 14. PMID 30224199